CLINICAL TRIAL: NCT02440568
Title: AML-02: Study of the Activity and Safety of the Addition of Omacetaxine to the Standard-of-Care Induction Therapy Regimen of Cytarabine and Idarubicin in Newly-Diagnosed AML Patients
Brief Title: AML-02: Omacetaxine With Standard-of-Care Induction With Cytarabine & Idarubicin in Newly-Diagnosed AML Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, John Quigley, Principal Investigator, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0181; 2015-0181 (Other: University of Illinois at Chicago)
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- Cohort 1: Omacetaxine at Dose level at 0.625mg/m^2 (Experimental): Patients will receive Omacetaxine at Dose level 0.625mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Omacetaxine mepesuccinate
- Cohort 2: Omacetaxine at Dose level at 1.25mg/m^ (Experimental): Patients will receive Omacetaxine at Dose level 1.25mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Omacetaxine mepesuccinate
- Cohort 3: Omacetaxine at Dose level at 2.0mg/m^ (Experimental): Patients will receive Omacetaxine at Dose level 2.0mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Omacetaxine mepesuccinate
- Cohort 4: Omacetaxine at Dose level at 3.0mg/m^ (Experimental): Patients will receive Omacetaxine at Dose level 3.0mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Interventions: Drug: Cytarabine; Drug: Idarubicin; Drug: Omacetaxine mepesuccinate

INTERVENTIONS:
Drug: Cytarabine — Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Other Names: Cytosine arabinoside, Ara-C, Cytosar
Drug: Idarubicin — Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
  Other Names: Idamycin PFS, Idamycin®
Drug: Omacetaxine mepesuccinate — Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Dose level 0.625mg/m^2
  Arms: Cohort 1: Omacetaxine at Dose level at 0.625mg/m^2
Drug: Omacetaxine mepesuccinate — Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Dose level 1.25mg/m^2
  Arms: Cohort 2: Omacetaxine at Dose level at 1.25mg/m^
Drug: Omacetaxine mepesuccinate — Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Dose level 2.0mg/m^2
  Arms: Cohort 3: Omacetaxine at Dose level at 2.0mg/m^
Drug: Omacetaxine mepesuccinate — Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Dose level 3.0mg/m^2
  Arms: Cohort 4: Omacetaxine at Dose level at 3.0mg/m^

SUMMARY:
This is a dose escalation study to evaluate Omacetaxine when given in combination with a standard induction regimen of "7+3" (cytarabine for Days 1-7 and Idarubicin for Days 1-3) in patients with newly diagnosed acute myelogenous leukemia (AML).

DETAILED DESCRIPTION:
This is a dose escalation study to evaluate Omacetaxine when given in combination with a standard induction regimen of "7+3" (cytarabine for Days 1-7 and Idarubicin for Days 1-3) in patients with newly diagnosed acute myelogenous leukemia (AML). Omacetaxine will be given subcutaneously Q12 hours on Days 1-7. The optimally safe and active dose (OD) will be determined using the EffTox design. EffTox is a Bayesian adaptive design that seeks to determine the optimal dose for further study in Phase II by considering a trade-off between efficacy and toxicity. The EffTox design begins by treating a cohort of three patients at dose level 1. These patients' efficacy and toxicity outcomes are used to update the posterior distributions for the probability of efficacy and toxicity and identify acceptable dose levels. The study terminates if no dose levels are acceptable. Otherwise, the acceptable doses are ranked using the Euclidean distance from (1.0, 0.0) and the next cohort is treated at the dose with the minimum distance under the restriction that we may only escalate or deescalate by one dose level at a time (e.g., the second cohort can only escalate to dose level 2 or deescalate to dose level -1). The second cohort is treated at the dose with the minimum distance and posterior distributions, and the list of acceptable doses and distances are updated as before. This process continues until at least 20 subjects are enrolled in the study. The dose with the minimum distance at study completion is considered the optimal dose for further investigation. If none of the dose levels are acceptable at study completion, an optimal dose level will not be identified and the drug does not warrant further investigation.

Post induction therapy will consist of standard cytarabine consolidation chemotherapy or allogeneic stem cell transplantation based on pretreatment risk assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, untreated patients with AML according to the WHO classification for AML. Prior short-term therapy (≤7 days) with hydroxyurea, steroids, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors, azacitidine, ATRA), or hematopoietic growth factors is allowed. A single or two-day dose of cytarabine (up to 3 g/m^2) for emergency use is also allowed as prior therapy.
2. Patients age 18 to 70 years old who meet diagnostic criteria for AML according to the WHO classification for AML.
3. Previously untreated AML (≥20% blasts). Note that prior short-term therapy (≤7 days) with hydroxyurea, steroids, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors, azacitidine, ATRA), or hematopoietic growth factors is allowed. A single or two-day dose of cytarabine (up to 3 g/m2) for emergency use is also allowed as prior therapy.
4. ECOG performance status of 0-3
5. Adequate organ function, if not suspected to be due to AML, within 14 days of study registration, defined as:

   Total bilirubin ≤ 2.0 x ULN (unless due to hemolysis) AST and ALT ≤ 3 X ULN (unless believed to be due to tumor involvement) Serum Creatinine ≤ 1.5 x ULN Creatinine Clearance > 30 ml/min
6. Negative urine or serum pregnancy test in females. Patients of reproductive potential (males and females) must consent to and practice double-barrier methods of contraception during treatment and for 12 weeks following the last dose of Omacetaxine. Adequate contraception is defined as double-barrier protection (i.e., condom plus spermicide in combination with a diaphragm, cervical/vault cap, or intrauterine device). Birth control pills, birth control patches and/or injections of hormones to prevent pregnancy are not considered an adequate method of preventing pregnancy, and double-barrier protection is required while on study and for 12 weeks after last dose. Patients will be instructed to notify the investigator if pregnancy is discovered either during or within 12 weeks of completing treatment with Omacetaxine. This also applies to male patients whose partners become pregnant while the patient is on study or within the 12 week period after the last dose of study drug.
7. Patients must be willing and able to review, understand, and provide written consent before starting therapy.

Exclusion Criteria:

1. Acute promyelocytic leukemia.
2. Investigational drug within 4 weeks of study entry.
3. Cardiac insufficiency grade III or IV New York Heart Association (NYHA)
4. Female subjects who are pregnant or breast feeding.
5. Patients who are HIV positive.
6. Active uncontrolled infection or severe systemic infection (enrollment is possible after control of infection).
7. Concurrent malignancy (other than AML) with an estimated life expectancy less than two years and requiring active therapy.
8. Psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up.
9. Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or medically relevant active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
10. Pregnant or breastfeeding: Omacetaxine is a Pregnancy Category D medication and has caused embryo-fetal death in animals. Confirmation that the subject is not pregnant must be established by a negative urine β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
11. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Quigley, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Newly Diagnosed AML, Cohort 1: Patients will receive Omacetaxine 0.625mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
- Patients With Newly Diagnosed AML, Cohort 2: Patients will receive Omacetaxine 1.25mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
- Patients With Newly Diagnosed AML, Cohort 3: Patients will receive Omacetaxine 2.0mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
- Patients With Newly Diagnosed AML, Cohort 4: Patients will receive Omacetaxine 3.0mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
Period: Overall Study
Arm/Group | Patients With Newly Diagnosed AML, Cohort 1 | Patients With Newly Diagnosed AML, Cohort 2 | Patients With Newly Diagnosed AML, Cohort 3 | Patients With Newly Diagnosed AML, Cohort 4
Started | 5 | 4 | 10 | 3
Completed | 1 | 1 | 5 | 1
Not Completed | 4 | 3 | 5 | 2
Not completed — Death | 1 | 3 | 4 | 2
Not completed — Lack of Efficacy | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Newly Diagnosed AML Cohort 1: Patients will receive Omacetaxine 0.625mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine (at assigned dose level) administered subcutaneously Q12 hours Days 1 to 7. Dose levels include: 0.625, 1.25, 2.0, 3.0, and 4.2 mg/m^2
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
- Patients With Newly Diagnosed AML Cohort 2: Patients will receive Omacetaxine 1.25mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine (at assigned dose level) administered subcutaneously Q12 hours Days 1 to 7. Dose levels include: 0.625, 1.25, 2.0, 3.0, and 4.2 mg/m^2
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
- Patients With Newly Diagnosed AML Cohort 3: Patients will receive Omacetaxine 2.0mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine (at assigned dose level) administered subcutaneously Q12 hours Days 1 to 7. Dose levels include: 0.625, 1.25, 2.0, 3.0, and 4.2 mg/m^2
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
- Patients With Newly Diagnosed AML Cohort 4: Patients will receive Omacetaxine 3.0mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine (at assigned dose level) administered subcutaneously Q12 hours Days 1 to 7. Dose levels include: 0.625, 1.25, 2.0, 3.0, and 4.2 mg/m^2
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
- Total: Total of all reporting groups
Arm/Group | Patients With Newly Diagnosed AML Cohort 1 | Patients With Newly Diagnosed AML Cohort 2 | Patients With Newly Diagnosed AML Cohort 3 | Patients With Newly Diagnosed AML Cohort 4 | Total
Number analyzed (Participants) | 5 | 4 | 10 | 3 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 7 | 2 | 18
  >=65 years | 0 | 0 | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 7 | 2 | 13
  Male | 3 | 2 | 3 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 4 | 0 | 6
  Not Hispanic or Latino | 4 | 3 | 6 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 1 | 6
  White | 2 | 3 | 7 | 2 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 10 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Optimally Tolerated Dose
Description: The primary endpoint is determination of the optimally active and safe dose (OD) of Omacetaxine when added to the standard-of-care induction chemotherapy for AML and estimation of the efficacy and response rate.
  OD will be defined as a dose level at which fewer than 30% of patients experience hematologic toxicity and greater than 50% of patients achieve a CR (50% is an accepted CR rate in AML when using a single induction).
Time Frame: Within 50 days (duration of hematologic recovery)
Population: Number of participants in each cohort
Measure: Number; unit: Participants treated with OD
Groups:
- Patients With Newly Diagnosed AML, Cohort 1: Patients will receive Omacetaxine 0.625mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
- Patients With Newly Diagnosed AML, Cohort 2: Patients will receive Omacetaxine 1.25mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
- Patients With Newly Diagnosed AML, Cohort 3: Patients will receive Omacetaxine 2.0mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
- Patients With Newly Diagnosed AML, Cohort 4: Patients will receive Omacetaxine 3.0mg/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
Arm/Group | Patients With Newly Diagnosed AML, Cohort 1 | Patients With Newly Diagnosed AML, Cohort 2 | Patients With Newly Diagnosed AML, Cohort 3 | Patients With Newly Diagnosed AML, Cohort 4
Number analyzed (Participants) | 5 | 4 | 10 | 3
Participants treated with OD | 0 | 0 | 10 | 0

2. Secondary Outcome: Toxicity: Describe by the Adverse Events as Assessed by the CTCAE Grading
Description: Describe the adverse events associated with Omacetaxine when administered in combination with cytarabine and Idarubicin as induction therapy for AML, using CTCAE grading
Time Frame: Up to 6 months after last dose of Omacetaxine
Population: All patients enrolled into the study
Measure: Number; unit: Total Adverse Events
Arm/Group | Patients With Newly Diagnosed AML, Cohort 1 | Patients With Newly Diagnosed AML, Cohort 2 | Patients With Newly Diagnosed AML, Cohort 3 | Patients With Newly Diagnosed AML, Cohort 4
Number analyzed (Participants) | 5 | 4 | 10 | 3
Total Adverse Events | 47 | 88 | 219 | 37

3. Secondary Outcome: Time to Hematologic Recovery
Description: Time to Absolute Neutrophil Count > 1.0 x 10e9/L and Platelet Count > 100 x 10e9/L, whichever was later, for those patients who achieved a remission and achieved these hematologic goals.
Time Frame: Within 6 months of last dose of Omacetaxine
Population: Patients who achieved a CR/CRi when treated with the study medications.
Measure: Median (Full Range); unit: Days
Groups:
- Patients With Newly Diagnosed AML, Cohort 3: Patients will receive Omacetaxine 2.0g/m^2, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine: Omacetaxine administered subcutaneously Q12 hours Days 1 to 7. Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
Arm/Group | Patients With Newly Diagnosed AML, Cohort 1 | Patients With Newly Diagnosed AML, Cohort 2 | Patients With Newly Diagnosed AML, Cohort 3 | Patients With Newly Diagnosed AML, Cohort 4
Number analyzed (Participants) | 2 | 3 | 4 | 1
Days | 25.5 [24 to 27] | 35 [24 to 37] | 33.5 [25 to 40] | 36 [36 to 36]

4. Secondary Outcome: Overall Participant Survival
Description: Observed overall survival among participants (days)
Time Frame: 3 years
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Patients With Newly Diagnosed AML, Cohort 1 | Patients With Newly Diagnosed AML, Cohort 2 | Patients With Newly Diagnosed AML, Cohort 3 | Patients With Newly Diagnosed AML, Cohort 4
Number analyzed (Participants) | 5 | 4 | 10 | 3
Days | 726 [360.5 to NA] — Insufficient number of participants with events | 162.5 [108 to NA] — Insufficient number of participants with events | 792.5 [91 to NA] — Insufficient number of participants with events | 33 [NA to NA] — Cannot calculate IQR on 3 participants

5. Secondary Outcome: Event Free Survival
Description: Observed length of time (days) after which patients remained free of recurrence or death.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Patients With Newly Diagnosed AML, Cohort 1 | Patients With Newly Diagnosed AML, Cohort 2 | Patients With Newly Diagnosed AML, Cohort 3 | Patients With Newly Diagnosed AML, Cohort 4
Number analyzed (Participants) | 5 | 4 | 10 | 3
Days | 66 [26.5 to NA] — Insufficient number of participants with events | 90.5 [50 to NA] — Insufficient number of participants with events | 65.5 [32 to NA] — Insufficient number of participants with events | 33 [NA to NA] — Cannot calculate IQR with 3 participants

6. Secondary Outcome: Progression Free Survival
Description: Among the participants who achieved CR,CRi, progression free survival in number of days, i.e. the number of days participants who achieved CR/CRi remained alive and in a remission.
Time Frame: 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Patients With Newly Diagnosed AML, Cohort 1 | Patients With Newly Diagnosed AML, Cohort 2 | Patients With Newly Diagnosed AML, Cohort 3 | Patients With Newly Diagnosed AML, Cohort 4
Number analyzed (Participants) | 2 | 3 | 4 | 1
Days | 852.5 [66 to 1639] | 100 [81 to 1480] | 1241.5 [793 to 1422] | 1141 [1141 to 1141]

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed for 1 year
Description: All-Cause Mortality was assessed for 3 years
Groups:
- Patients With Newly Diagnosed AML, Cohort 1: Patients will receive Omacetaxine, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine at Dose level at 0.625mg/m^2 administered subcutaneously Q12 hours Days 1 to 7.
  Cytarabine: Cytarabine (100mg/m^2/day) in 1000ml NS as a continuous IV infusion over 24 hours x 7 days.
  Idarubicin: Idarubicin (12 mg/m^2/day) IVPB in 100 mL NS over 15 minutes daily from Days 1 to 3.
- Patients With Newly Diagnosed AML, Cohort 2: Patients will receive Omacetaxine, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine at Dose level at 1.25mg/m^2 administered
- Patients With Newly Diagnosed AML, Cohort 3: Patients will receive Omacetaxine, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine at Dose level at 2.0mg/m^2 administered
- Patients With Newly Diagnosed AML, Cohort 4: Patients will receive Omacetaxine, Cytarabine and Idarubicin as part of the treatment plan. Study participants will follow in outpatient clinic at least every 2 months for a total of 6 months. A final study visit will occur 6 months (+/-1 week) after the last dose of Omacetaxine. This visit will end study participation unless there is ongoing toxicity that is at least possibly related to study treatment. In this case, the patient will be followed as medically appropriate until resolution or stabilization of the adverse event.
  Omacetaxine at Dose level at 3.0mg/m^2 administered
Arm/Group | Patients With Newly Diagnosed AML, Cohort 1 | Patients With Newly Diagnosed AML, Cohort 2 | Patients With Newly Diagnosed AML, Cohort 3 | Patients With Newly Diagnosed AML, Cohort 4
All-Cause Mortality (participants affected / at risk) | 2/5 | 3/4 | 4/10 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/4 | 4/10 | 2/3
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 10/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Newly Diagnosed AML, Cohort 1 (N=5) | Patients With Newly Diagnosed AML, Cohort 2 (N=4) | Patients With Newly Diagnosed AML, Cohort 3 (N=10) | Patients With Newly Diagnosed AML, Cohort 4 (N=3)
Death (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2) — Progression of disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Newly Diagnosed AML, Cohort 1 (N=5) | Patients With Newly Diagnosed AML, Cohort 2 (N=4) | Patients With Newly Diagnosed AML, Cohort 3 (N=10) | Patients With Newly Diagnosed AML, Cohort 4 (N=3)
Chills (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Infusion related reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiorgan failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Weight loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypervolemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Edema to lims (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Facial edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Oral mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascities (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Epistaxis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acute coronary syndrom (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 9 (9) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Septic emboli (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Esophageal infection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vulvlar abscess (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypophosphemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Increased alkaline phosphatse (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Increased alanine aminotransferase (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Increased aspartate aminotransferase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased blood bilirubin (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Increased INR (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Increased PTT (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Decreased urinary output (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloody stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastric bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Delirium (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rentinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT02440568/Prot_SAP_000.pdf